CLINICAL TRIAL: NCT07192133
Title: Evaluation of Computed Tomography X-ray-Pulsatility Index (CT-XPI)
Brief Title: Evaluation of CT-XPI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-0586; SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); AS (Other: UW Madison); Protocol Version 1/18/2025 (Other: UW Madison)
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: CT Scan; Computed Tomography
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CT scan (Experimental): Participants undergoing a CT
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — Dynamic contrast-free chest CT scan

SUMMARY:
The goal of this clinical trial is to learn if a new computed tomography (CT) lung perfusion imaging method is as effective as standard of care (SOC) CT imaging. The main question it aims to answer is:

* Does the new contrast-free method provide more information about lung perfusion than SOC?

Participants will undergo a 30 minute chest CT.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate X-ray Pulsatility Index using prospectively acquired dynamic CT, which is different from conventional static CT scans.

The primary objective of this study is to collect dynamic CT scan data with human participants using high frame rate imaging methods to produce a map of lung perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to sign and date the informed consent form
* Will undergo a clinically-indicated CT exam of the head, neck, chest, abdomen, pelvis, or extremities

Exclusion Criteria:

* Pregnant or lactating
* In need of urgent or emergent care
* Have any conditions that, in the opinion of the PI or designee, would interfere with the evaluation of the results or constitute a health hazard for the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lung x-ray pulsatility index (XPI) | 30 minutes
  XPI, a representative of lung perfusion, will be measured using CT images. The dynamic x-ray attenuation from each pixel is analyzed using spectral analysis.
Magnitude of XPI | 30 minutes
  Measured as a number, this corresponds to the magnitude of the relative change of signal.
Presence of XPI | 30 minutes
  This will be evaluated quantitatively using CNR (contrast to noise) measurements which uses a region of interest in the lungs and a region of interest outside of the lungs.
Spatial distribution of XPI signal | 30 minutes
  This is a subjective evaluation, routinely done clinically with other modalities that measure lung perfusion. Researchers evaluate how homogenous (smooth) the signal is over the lungs and look for perfusion defects (areas with little or no XPI) which would indicate pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes